CLINICAL TRIAL: NCT07143604
Title: A Phase II, Multicentre, Open-label, Single-arm Study of AZD0901 Monotherapy in Second-or Later-Lines Adult Participants With Advanced/Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Expressing Claudin18.2
Brief Title: A Study to Investigate the Effects of AZD0901 Monotherapy in Adult Participants With 2L+ Advanced or Metastatic Gastric or GEJ Adenocarcinoma Expressing CLDN18.2
Acronym: GAMBIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-RU-00007
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Gastric cancer; Gastroesophageal junction cancer; Claudin 18.2; AZD0901
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will receive AZD0901 IV, Q3W
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD0901 (Experimental): Participants will receive AZD0901 IV, Q3W
  Interventions: Drug: AZD0901

INTERVENTIONS:
Drug: AZD0901 — Participants will receive AZD0901 IV, Q3W
  Other Names: Sonesitatug Vedotin

SUMMARY:
The purpose of this study is to measure the efficacy and safety of AZD0901 monotherapy as 2L+ treatment for participants with advanced or metastatic gastric or GEJ adenocarcinoma expressing CLDN18.2.

DETAILED DESCRIPTION:
This is a Phase II, single arm, open label, multicentre study, assessing the efficacy and safety of AZD0901 in participants with advanced/metastatic gastric or gastroesophageal junction adenocarcinoma expressing Claudin18.2. The results of the study will provide clinical data on efficacy and safety of an innovation drug in Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of gastric, GEJ, or distal esophagus, with positive CLDN18.2 expression.
* Disease progression on or after at least one prior regimen for advanced or metastatic disease, which included a fluoropyrimidine and a platinum, for advanced or metastatic disease.
* Must have at least one measurable lesion assessed by the Investigator based on RECIST 1.1.
* ECOG performance status of 0 or 1.
* Minimum life expectancy of ≥12 weeks.
* Adequate organ and bone marrow function.
* Minimum body weight of 40 kg.
* Sex and Contraceptive Requirements.

Exclusion Criteria:

* Participants with known HER2 positive status as defined as IHC 3+ or IHC 2+/ISH +.
* Participant has significant or unstable gastric bleeding and/or untreated gastric ulcers.
* CNS metastases or CNS pathology.
* Participant has known clinically significant corneal disease (eg, active keratitis or corneal ulcerations).
* Persistent toxicities (CTCAE Grade ≥2) caused by previous anticancer therapy.
* History of thromboembolic events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At month 6 after date of first dose
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, as determined by the investigator per RECIST 1.1 to all dosed participants

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 30 months
  PFS is defined as time from date of first dose until progression per RECIST 1.1 as assessed by the investigator, or death due to any cause
Overall Survival (OS) | From the date of assignment until the date of death from any cause, assessed up to 30 months
  OS is defined as the time from date of first dose of IMP until the date of death due to any cause. The analysis will include all dosed participants. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy
Disease control rate (DCR) at 12 weeks | At 12 weeks after date of first dose
  DCR at 12 weeks is defined as the percentage of participants who have at least 1 visit response of confirmed CR or PR or who have stable disease (SD) per RECIST 1.1 for at least 11 weeks as assessed by the investigator to all dosed participants
Duration of Response (DoR) | From the date of first documented confirmed response until date of documented progression, assessed up to 30 months
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression or death due to any cause. Analysis will include all dosed participants, with measurable disease at baseline who have a response, regardless of whether the participant withdraws from therapy, receives another anticancer treatment, or clinically progresses prior to PD.
Time to Response (TTR) | From the date of first dose to the first documented objective tumor response, assessed up to 30 months
  TTR is defined as the time from the start of the treatment to the first documented objective tumor response observed for participants who achieved CR or PR, as determined by the investigator according to RECIST 1.1. Analysis will include all dosed participants, with measurable disease at baseline who have a response, regardless of whether the participant withdraws from therapy, receives another anticancer treatment, or clinically progresses prior to PD.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | From the time of ICF signature up to 30 months
  Treatment-emergent adverse events are defined as adverse events or worsening of pre-existing events with an onset date on or after first dose of IMP and within 90 (+ 7) days after last dose of study intervention or up to the day prior to start of subsequent therapy, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Research Site, Chelyabinsk
  - Research Site, Krasnoyarsk
  - Research Site, Kuzmolovskiy
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Volgograd

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home